CLINICAL TRIAL: NCT04877041
Title: Trial of Intradialytic Cycling as Kidney Exercise Rehabilitation for Cardiac Stunning in Hemodialysis (TICKERS-HD)
Brief Title: Exercise and Cardiac Stunning During HD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS24857 (B2021:039)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: End-stage Kidney Disease; Hemodialysis
Keywords: intradialytic exercise
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts will also be blinded to study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Intradialytic Cycling) (Experimental): Participants will receive a standardized baseline exercise counseling session as per control and then participate in a supervised intradialytic cycling program for 12-weeks
  Interventions: Behavioral: Intradialytic Cycling
- Usual Care (No Intervention): Participants will receive a standardized baseline exercise counseling session. Participants in the control group will not undergo formal exercise intervention, but will not be prohibited from participating in exercise outside of hemodialysis. They will be asked to not to participate in intradialytic cycling during the study (16 weeks total).

INTERVENTIONS:
Behavioral: Intradialytic Cycling — This intervention will consist of intradialytic cycling for 60 minutes 3 times per week for a total of 12 weeks.
  Arms: Exercise (Intradialytic Cycling)

SUMMARY:
The purpose of this study is to determine the effect of a 12-week cycling during hemodialysis program on hemodialysis-induced myocardial stunning in adult individuals receiving hemodialysis.

DETAILED DESCRIPTION:
People with kidney failure receiving chronic hemodialysis (HD) suffer from post-HD treatment fatigue, poor functional status and high rates of cardiac failure and death. Previous work has shown that these outcomes are correlated with recurrent ischemic cardiac injury (myocardial stunning) that occurs during HD treatments. Myocardial stunning, identified by regional cardiac wall motion abnormalities (RWMA), is common during HD. Intradialytic cycling (during HD) decreases HD-induced stunning, and may improve adverse outcomes associated with stunning. We will use echocardiography (echo) to understand the effects of intradialytic aerobic exercise on myocardial stunning and HD-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years old (no upper age limit); who are greater than; 3 months after starting maintenance hemodialysis
* No expected change in dialysis modality, elective surgery or relocation outside of study site during the intervention period (16 weeks)
* Assessed to be safe and able to exercise by the hemodialysis unit nephrologist
* Able to communicate in English and provide written informed consent
* Must be dialyzing thrice weekly

Exclusion Criteria:

* Acute coronary syndrome in the past 3 months
* Unstable arrhythmia
* Shortness of breath at rest or with minimal activity (NYHA Class 4)
* Symptomatic hypoglycemia (>2x/week in week prior to enrolment)
* Participating in clinical intradialytic cycling program in last 3 months (if a clinical program exists)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in number of cardiac RWMA at peak hemodialysis stress (last 30 min HD) from baseline to 12 weeks measured using echocardiography | Baseline to 12 weeks
  Using standard left ventricular apical 2-, 3-, and 4-chamber views and left ventricular parasternal short-axis views collected by the same trained operator at each site 3 times during the mid-week hemodialysis session at each assessment time point as follows: baseline (pre hemodialysis), post-cycling exercise (or mid-dialysis in controls) and at peak hemodialysis stress (~30 min prior to end of hemodialysis). Echocardiogram image analysis will be performed in London, ON using automated speckle-tracking analysis (EchoPAC-PC software version 110.1.3; GE Healthcare).

SECONDARY OUTCOMES:
Change in post-hemodialysis high sensitivity Troponin T level from baseline to 12 weeks | Baseline to 12 weeks
  Measured by Roche High-Sensitivity Troponin T assay at each site.
Change in difference between pre-hemodialysis and post-hemodialysis Troponin T from baseline to 12 weeks | Baseline to 12 weeks
  Measured by Roche High-Sensitivity Troponin T assay at each site.
Change in number of cardiac RWMA at peak hemodialysis stress (last 30 min HD) from baseline to 16 weeks measured using echocardiography | Baseline to 16 weeks
  Using standard left ventricular apical 2-, 3-, and 4-chamber views and left ventricular parasternal short-axis views collected by the same trained operator at each site 3 times during the mid-week hemodialysis session at each assessment time point as follows: baseline (pre hemodialysis), post-cycling exercise (or mid-dialysis in controls) and at peak hemodialysis stress (~30 min prior to end of hemodialysis). Echocardiogram image analysis will be performed in London, ON using automated speckle-tracking analysis (EchoPAC-PC software version 110.1.3; GE Healthcare).
Change in severity of post-hemodialysis fatigue | Baseline to 12 weeks
  Assessed by the self-reported answer (in minutes) to the question: "How long does it take you to recover from a dialysis session and resume your normal, usual activities?"
Change in Symptom Burden | Baseline to 12 weeks
  Measured using the Dialysis Symptom Index (DSI) Severity Score. Score 0 to 150 with 0 no symptoms and 150 most number and severity of symptoms
Change in Exercise Capacity | Baseline to 12 weeks
  Measured by the Incremental Shuttle Walk Test (ISWT)
Change in Physical Activity Behaviour Patterns | Baseline to 12 weeks
  Assessed using total active minutes per day as measure by multi-directional accelerometry
Change in number of regional wall motion abnormalities at peak HD stress | Baseline to 1 week
  Measured at each study time point to further assess how exercise training effects HD-related cardiac stunning over time
Change in number of regional wall motion abnormalities at peak HD stress | Baseline to 16 weeks
  Measured at each study time point to further assess how exercise training effects HD-related cardiac stunning over time
Feasiblity - Recruitment | Baseline to 12 weeks
  Proportion of individuals eligible for study that were recruited
Feasibility - Eligibility | Baseline to 12 weeks
  Proportion of individuals approached eligible for enrolment into study
Feasibility - Adherence | Baseline to 16 weeks
  Proportion of participants that completed the study
Feasibility - Exercise Adherence: Proportion of exercise sessions completed | Baseline to 12 weeks
  Proportion of total exercise sessions during study completed
Feasibility - Exercise Adherence: Total minutes of exercise | Baseline to 12 weeks
  Proportion of total possible minutes of intradialytic cycling completed during the study
Change in Cognitive Function | Baseline to 12 weeks
  Change in cognitive function score measured by Cambridge Brain Science testing
Change in number of cardiac RWMA at peak hemodialysis stress (last 30 min HD) from 12 to 16 weeks measured using echocardiography | From 12 to 16 weeks
  Using standard left ventricular apical 2-, 3-, and 4-chamber views and left ventricular parasternal short-axis views collected by the same trained operator at each site 3 times during the mid-week hemodialysis session at each assessment time point as follows: baseline (pre hemodialysis), post-cycling exercise (or mid-dialysis in controls) and at peak hemodialysis stress (~30 min prior to end of hemodialysis). Echocardiogram image analysis will be performed in London, ON using automated speckle-tracking analysis (EchoPAC-PC software version 110.1.3; GE Healthcare).

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bohm, MD, MPH, Principal Investigator — University of Manitoba
Locations (6):
- University of South Australia, Adelaide, South Australia, Australia
- Canada (5):
  - University of Calgary Cumming School of Medicine Department of Internal Medicine, Calgary, Alberta
  - University of Alberta Department of Internal Medicine, Edmonton, Alberta
  - St. Pauls Hospital, Vancouver, British Columbia
  - University of Manitoba Department of Internal Medicine, Winnipeg, Manitoba
  - Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett PN, Penny JD, McIntyre CW, Vanderlinden J, Borkum MS, Castillo G, Collister D, Corradetti B, Duhamel TA, Farion H, Ford E, Garcia E, Getachew R, Jesudason S, Kiaii M, Leu RL, Presseau J, Rigatto C, Seitz AK, Shirazi M, Soni A, Stewart K, Tarca B, Tennankore K, Verdin N, Whitlock R, Wilund K, Thompson S, MacRae JM, Bohm C. Randomized Controlled Trial of Intradialytic Cycling as Kidney Exercise Rehabilitation for Cardiac Stunning in Hemodialysis (TICKERS_HD): A Clinical Research Protocol. Can J Kidney Health Dis. 2026 Jan 17;13:20543581251391112. doi: 10.1177/20543581251391112. eCollection 2026. PMID 41555861
- [Derived] McIntyre CW. Update on Hemodialysis-Induced Multiorgan Ischemia: Brains and Beyond. J Am Soc Nephrol. 2024 May 1;35(5):653-664. doi: 10.1681/ASN.0000000000000299. Epub 2024 Jan 26. PMID 38273436